CLINICAL TRIAL: NCT04515368
Title: A Pilot Clinical Study of PET Scanning in Evaluation of Vaccine Reactogenicity
Acronym: PETVACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PETVACC; 15/LO/2039 (Other: London 'Äì Surrey Borders Research Ethics Committee); 191407 (Other: IRAS project ID)
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Positron-Emission Tomography; Immunization Reaction
MeSH Terms: interventions — Immunization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fendrix (Experimental): Fendrix (Hepatitis B surface antigen adjuvanted by AS04C containing 3¬≠O¬≠desacyl¬≠4'¬≠ monophosphoryl lipid A adsorbed on aluminium phosphate, GlaxoSmithKline; 0.5 mL. intramuscular. stat.
  Interventions: Biological: Immunization
- Bexsero (Experimental): Bexsero (Meningococcal group B subunit / Outer Membrane Vesicles, GlaxoSmithKline); 0.5 mL. intramuscular. stat.
  Interventions: Biological: Immunization
- Fluad (Experimental): Fluad (split virion inactivated seasonal trivalent influenza vaccine adjuvanted with MF59C, Northern Hemisphere 2016-17, Seqirus Vaccines and Diagnostics) 0.5 mL. intramuscular. stat.
  Interventions: Biological: Immunization
- Seasonal Trivalent Influenza Vaccine (Experimental): Seasonal Trivalent Influenza Vaccine ('ÄòSTIV'Äô, split virion inactivated, Northern Hemisphere 2016-17, Sanofi Pasteur); 0.5 mL. intramuscular. stat.
  Interventions: Biological: Immunization

INTERVENTIONS:
Biological: Immunization — Immunisation with one of four licensed vaccines

SUMMARY:
This study forms part of an integrated, multi-study effort to identify potential biomarkers of reactogenicity to vaccines. We have selected PET-CT as it is in routine clinical use and has been serendipitously shown to image lymph nodes and injection site inflammation after immunisation.The study's objectives are exploratory:

1. To methodically characterise relative anatomical distribution and intensity of post-immunisation innate immune activation visualised by PET-CT after immunisation with adjuvanted and non-adjuvanted vaccines.
2. To correlate PET/CT changes with diary card recorded symptoms of reactogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read and understand the informed consent form (ICF), and understand study procedures
2. Signed the ICF
3. Healthy male aged 18'Äì55 years inclusive
4. BMI 19'Äì27 kg/m2
5. Pre-immunised with hepatitis B vaccine on the basis of immunisation history if Fendrix or Engerix B is to be the study vaccine
6. Available for follow-up for the duration of the study
7. Is, in the opinion of the investigator, healthy on the basis of a medical history, symptom directed medical examination and vital signs
8. Have not undergone research radiation exposures, and agree to avoid such exposures, for 12 months before/after this study
9. Be willing to avoid vigorous exercise or contact sports between vaccination and PET scan (e.g. gym workouts, prolonged cycling, rowing, martial arts or rugby)

Exclusion Criteria:

1. History of hypersensitivity to any of the vaccine components or a history of any allergy that in the opinion of the investigator would contraindicate participant participation
2. Use of steroids or immunosuppressive/immunomodulating drugs either orally or parenterally within 3 months of the PET scan. (Topical/ocular/nasal/inhaled steroids are allowed.)
3. Expression of only TSPO with low-affinity to PBR28, on the basis of TSPO genotype
4. Currently participating in a clinical study with a drug or device
5. Any condition that, in the investigator'Äôs opinion, compromises the participant'Äôs ability to meet protocol requirements or to complete the study
6. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
18FDG-PET/CT imaging | 4 hours
  Quantification of PET activity at injection site and draining lymph nodes
18FDG- or 11C-PBR28-PET/CT imaging | 1 day
  Quantification of PET activity at injection site and draining lymph nodes
18FDG- or 11C-PBR28-PET/CT imaging | 3 days
  Quantification of PET activity at injection site and draining lymph nodes
18FDG- or 11C-PBR28-PET/CT imaging | 5 days
  Quantification of PET activity at injection site and draining lymph nodes
18FDG- or 11C-PBR28-PET/CT imaging | 7 days
  Quantification of PET activity at injection site and draining lymph nodes
18FDG-PET/CT imaging | 10 days
  Quantification of PET activity at injection site and draining lymph nodes

SECONDARY OUTCOMES:
Diary card of reactogenicity | 0 to 10 days
  Recording of solicited and unsolicited adverse events after immunisation

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — Imperial College Healthcare NHS Trust

IPD SHARING:
Plan to Share IPD: No